CLINICAL TRIAL: NCT02438618
Title: Minimally Invasive Surgery for Ponto Bone Anchored Hearing Implants
Acronym: C50
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C50
Record Dates: First submitted 2015-04-21; First posted 2015-05-08 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Conductive Hearing Loss; Unilateral Partial Deafness; Mixed Conductive-sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimally invasive punch technique (Experimental): New surgical technique for Ponto bone anchored hearing implants
  Interventions: Procedure: Surgery for Ponto bone anchored hearing aids
- Hultcrantz technique (Other): Standard surgical technique for bone anchored hearing implants
  Interventions: Procedure: Surgery for Ponto bone anchored hearing aids

INTERVENTIONS:
Procedure: Surgery for Ponto bone anchored hearing aids

SUMMARY:
The objective of this study is to make a comparison between two surgical techniques used when implanting a Ponto bone anchored hearing system.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, i.e. ≥ 18 years of age
* Eligible for the Ponto system

Exclusion Criteria:

* Known history of immunosuppressive disease
* Use of systemic immunosuppressive medication
* Receiving bilateral bone anchored hearing system
* Relevant dermatological diseases as judged by the investigator
* Not being able to finish the study, for example because of failure to complete the questionnaires
* Participating in another study with medical aids or medication
* When there is no suitable implantation-site for the 4 mm implant during surgery because of insufficient bone quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2018-11-18 (Actual)

PRIMARY OUTCOMES:
Incidence of inflammation (Holgers index ≥ 2) | 3 months post surgery

SECONDARY OUTCOMES:
Presence of dehiscence after surgery (Noted in a binary fashion (present/not present)) | 3 months post surgery
Visual Analogue Scale (VAS) pain scale > 6 (Noted on a scale from 0 - 10) | 3 months post surgery
Loss of sensibility (Measured in mm outwards from the abutment) | 3 months post surgery
Soft tissue overgrowth (mm) | 3 months post surgery
Extrusion rate (number of implants lost) | 3 months post surgery
Implant stability quotient (ISQ) measurements (ISQ units 1-100) | 3 months post surgery
Surgical time (minutes) | 3 months post surgery
Wound healing time (time to reach healed) | 3 months post surgery
Holgers index ≥ 2 at any time point | 24 months post surgery
Presence of dehiscence after surgery (present/not present) | 24 months post surgery
Visual Analogue Scale (VAS) pain scale > 6 (Noted on a scale from 0 - 10) | 24 months post surgery
Loss of sensibility (Measured in mm outwards from the abutment) | 24 months post surgery
Soft tissue overgrowth (mm) | 24 months post surgery
Extrusion rate (number of implants lost) | 24 months post surgery
Implant stability quotient (ISQ) measurements (ISQ units 1-100) | 24 months post surgery
  Measured in ISQ units (1-100)
Cosmetic result (10 point scale) | 24 months post surgery
  Scored using a 10-point scale and are compared to the healthy, normal contralateral situation

OTHER OUTCOMES:
Skin position (analysed descriptively using photographs and computer software) | 3 months post surgery
  Only at main center
Dynamic skin motion (analysed descriptively using photographs and computer software) | 3 months post surgery
  Only at main center
Quality of life related questionnaires | 24 months post surgery
Correlation between cytokines and Holgers index | 24 months post surgery
Correlation IS-pro profile and Holgers index | 24 months post surgery
Development of a peri-implant dermatitis scale and compare it to the Holgers Index | 24 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stokroos, Professor, Principal Investigator — Maastricht University Medical Centre (MUMC+)
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Strijbos RM, Straatman LV, Stegeman I, Holmberg M, Johansson ML, Stokroos RJ. Health Economic Cost Analysis for Percutaneous Bone Conduction Devices: The Minimally Invasive Ponto Surgery Versus Linear Incision Technique with Tissue Preservation. Otol Neurotol. 2023 Aug 1;44(7):709-717. doi: 10.1097/MAO.0000000000003939. Epub 2023 Jun 29. PMID 37400140
- [Derived] Strijbos RM, Straatman LV, Calon TGA, Johansson ML, de Bruijn AJG, van den Berge H, Wagenaar M, Eichhorn E, Janssen M, Jonhede S, van Tongeren J, Holmberg M, Stokroos R. Long-Term Outcomes of the Minimally Invasive Ponto Surgery vs. Linear Incision Technique With Soft Tissue Preservation for Installation of Percutaneous Bone Conduction Devices. Front Neurol. 2021 Feb 24;12:632987. doi: 10.3389/fneur.2021.632987. eCollection 2021. PMID 33716934
- [Derived] Calon TG, van Hoof M, van den Berge H, de Bruijn AJ, van Tongeren J, Hof JR, Brunings JW, Jonhede S, Anteunis LJ, Janssen M, Joore MA, Holmberg M, Johansson ML, Stokroos RJ. Minimally Invasive Ponto Surgery compared to the linear incision technique without soft tissue reduction for bone conduction hearing implants: study protocol for a randomized controlled trial. Trials. 2016 Nov 9;17(1):540. doi: 10.1186/s13063-016-1662-0. PMID 27829464